CLINICAL TRIAL: NCT06236867
Title: The Effect of Ice Application and Kaleidoscope Application on the Management of Cannulation-Related Pain in Dialysis Patients With Arteriovenous Fistula
Brief Title: Cannulation-Related Pain in Dialysis Patients With Arteriovenous Fistula
Acronym: AVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sülayman YAMAN (Other)
Responsible Party: Sponsor-Investigator, Sülayman YAMAN, Master Student, Amasya University
Organization: Amasya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AU-SBE-SY-01
Record Dates: First submitted 2023-12-27; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hemodialysis Access
Keywords: Arteriovenous fistula; Nursing; Pain Management
MeSH Terms: conditions — Arteriovenous Fistula; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After obtaining the necessary permissions for the research, the patients who were followed up in the hemodialysis unit of X,Y, Z Hospitals were randomly divided into three groups (Kaleidoscope application, ice application and control group).
  Patients were made to sign written voluntary consent forms by the researchers.After the patients were transferred to the randomized program for the arrival days and TC numbers for the dialysis session, they were assigned to the experimental and control groups.
  The patients' pain levels were evaluated during 3 dialysis sessions. The pain level was evaluated without the procedure on the first day. 2 and 3. on the other hand, pain levels were evaluated after the interventions per day.
  The data in the research are; Patient Diagnosis Form, Numerical Rating Scale and Life Signs Follow-up Form and Kaleidoscope Application Patient Experience Form, It was collected using the Patient Experience Form Related to Ice Application.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients did the pain scoring without knowing which group they were in. Patients are blinded.
  In order to prevent the groups from being affected by each other, a inspection curtain was placed between the dialysis machines during the applications.
  The data were coded as A, B and C groups and sent for statistical analysis. The outcomes assesor doing the analysis here is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kaleidoscope Group (Experimental): In order for the patients in the kaleidoscope group to recognize the device and increase their compliance during the procedure, a practice was performed using the device before the AVF cannulation procedure. Kaleidoscope application was performed during cannulation.
  Interventions: Other: KaleidoscopeGroup
- Ice Application Group (Experimental): Ice application application was made with non-melting ice molds to the area where the index finger and thumb of the hand with fistula are joined (HOKU point).
  Interventions: Other: Ice Application Group
- Control Group (Experimental): In the control group, the vital signs of the patients before AVF cannulation will be recorded. Before, during and after AVF cannulation, VAS pain scores will be evaluated after cannulation without any intervention.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: KaleidoscopeGroup — The group consists of 34 people. Pain level was measured during 3 dialysis sessions.In order for the patients in the kaleidoscope group to recognize the device and increase their compliance during the procedure, a practice was performed using the device before the AVF cannulation procedure. Kaleidoscope application was performed during cannulation.
  Other Names: Experimental
  Arms: Kaleidoscope Group
Other: Ice Application Group — The group consists of 34 people. Pain level was measured during 3 dialysis sessions. Before, during and after AVF cannulation, VAS pain scores will be evaluated after cannulation without any intervention.Ice application application was made with non-melting ice molds to the area where the index finger and thumb of the hand with fistula are joined (HOKU point)
  Other Names: Experimental
  Arms: Ice Application Group
Other: Control Group — The group consists of 34 people. Pain level will be measured during 3 dialysis sessions. In the control group, the vital signs of the patients before AVF cannulation will be recorded.
  Other Names: Experimental
  Arms: Control Group

SUMMARY:
It was conducted to investigate the effect of ice application to the kaleidoscope and hoku point on the management of cannulization-related pain in patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
After obtaining the necessary permissions for the research, the patients who were followed up in the hemodialysis unit of X,Y, Z Hospitals were randomly divided into three groups (Kaleidoscope application, ice application and control group).

Patients were made to sign written voluntary consent forms by the researchers.After the patients were transferred to the randomized program for the arrival days and TC numbers for the dialysis session, they were assigned to the experimental and control groups.

The patients' pain levels were evaluated during 3 dialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

Comfortable reception of trill and murmur sound from arteriovenous fistula,

• over the age of 18 and no communication problems,

* Having a place and time orientation,
* No dizziness,

Exclusion Criteria:

* Hemodialysis of the patient with arteriovenous graft and/or central venous catheter
* Pharmacological application was made to relieve pain 30 minutes before AVF cannulation,

  * The patient has a COVID - 19 infection
  * Having visual, auditory and intellectual disabilities,
  * Having a communication problem,
  * Not willing and willing to participate in the study, as well as wanting to withdraw from the study at any stage of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Over age the 18
Enrollment: 102 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
visual pain scale (min-max:0-10 point) (1 week= during 3rd dialysis sessions) | One week= during 3rd dialysis sessions
  Evaluation of pain levels (minimum=0 points, maximum: 10 points) of experimental and control groups in the 1st, 2nd and 3rd dialysis sessions
  The visual pain scale is minimum 0 and maximum 10 points. 0 means no pain, 10 means severe pain.
  1. st dialysis session= Visual analog pain scores during cannulation were evaluated without any application.
  2. nd and 3rd dialysis sessions: Ice application to the patient's hoku point was performed by the researcher for 1 min before the AVF cannulation procedure and during cannulation, and visual analog scale pain scores was filled in during cannulation.
  Kaleidoscope application was performed to the patient for 5 minutes before AVF cannulation procedure and during cannulation. The visual analog scale pain score was filled in during cannulation.
  Control Group:visual analog scale pain scores will be evaluated before, during and after AVF cannulation without any intervention after the procedure.

SECONDARY OUTCOMES:
The evaluation of Ice Application and kaleidoscope application | After 3rd dialysis session (after one week)
  Learning patient experiences regarding ice application and kaleidoscope application via Kaleidoscope Application Patient Experience Form, Patient Experience Form for Ice Application.
  The answers of the participants to the questions in the evaluation forms (Kaleidoscope Application Patient Experience Form, Patient Experience Form for Ice Application) are presented as a percentage. They were asked to answer the questions asked in the form as "yes, no, partially".
Sociodemographic and disease-related characteristics | through study completion, an average of 3rd month.
  Comparison of sociodemographic characteristics (age, gender) with visual pain scale scores of the experimental and control groups.
  Comparison of disease-related characteristics [Body mass index:weight and height will be combined to report BMI in kg/m^2 (weight in kilograms, height in meters=kg/m2), duration of dialysis (months), artery and vein needle size (14,15,16,17 gauge), duration of fistula use, region where the fistula is located)] with visual pain scale scores of the experimental and control groups.
  NOTE:After the data in all dialysis centers were completed (within about three months), the analysis was performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University İnstitute of Health Sciences, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results will be shared when the author is requested for meta-analysis studies.